CLINICAL TRIAL: NCT04653948
Title: Prevention of Invasive Group B Streptococcus Disease in Young Infants: a Pathway for the Evaluation & Licensure of an Investigational Maternal GBS Vaccine (Work Package 2)
Brief Title: Maternal, Neonatal and Infant Outcomes at Kawempe National Referral Hospital
Acronym: PREPARE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Collaborators: MU-JHU CARE (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: 17.0020
Record Dates: First submitted 2020-11-10; First posted 2020-12-04 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Group B Streptococcus Carrier in Childbirth; Group B Streptococcal Infection, Late-Onset; Group B Streptococcal Infection, Early-Onset; Group B Streptococcus Neonatal Sepsis; Group B Strep Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort Study: Women greater than or equal (≥) to 18 years of age and emancipated minors aged between 14 and 17 years of age seeking antenatal care at Kawempe National Referral Hospital in their first and second trimesters of pregnancy will be invited to participate in the study until a sample size of at least 4000 women is achieved. They will be followed-up along with their liveborn infants until a minimum of 14 weeks post-delivery.
- EMR Cohort: Anonymised data from the entire maternal and infant population that attend Kawempe Hospital for antenatal and/or delivery +/- post-partum care during the two-year study period will be analysed to describe maternal, obstetric and neonatal outcomes.

SUMMARY:
Maternal immunisation is an evolving field that deserves special attention given its potential to have a significant positive impact on the health of women and children globally, and the potential safety and risk considerations associated with research in this population.

The goal of maternal immunisation is to boost maternal levels of specific antibodies to provide the newborn and young infant with sufficient immunity at birth, through trans placental transfer in-utero, to protect them through the period of increased vulnerability. Protection should be adequate to last until they are able to respond to their own active immunisations or infectious challenges. The success of the maternal neonatal tetanus immunisation program demonstrates the utility of this approach. Several other vaccines are recommended in pregnancy, including influenza and pneumococcal vaccines. Promising new vaccines for group B streptococcus (GBS) , respiratory syncytial virus (RSV) and cytomegalovirus are under development. They are targeted for use in pregnant women in high-, middle-, and low-income countries. However, these vaccines are likely to be of most benefit in LMICs that have high rates of vaccine preventable diseases.

The second work-package (WP2) of the PREPARE portfolio will describe the baseline maternal and neonatal outcomes using anonymised data collected using the routine Kawempe electronic medical records (EMR) system.

Furthermore, comprehensive data on pregnancy, neonatal and infant outcome will also be collected in a prospective cohort of women enrolled in the first and second trimesters while attending antenatal care at Kawempe Hospital with follow-up of the mother-infant pair(s) up until at least 14 weeks postpartum to establish longer term outcomes. Standardised case definitions will be used to classify the outcomes.

DETAILED DESCRIPTION:
Maternal Immunisation research in LMICs

Maternal immunisation is an evolving field that deserves special attention given its potential to have a significant positive impact on the health of women and children globally, and the potential safety and risk considerations associated with research in this population.

Prior to undertaking any maternal vaccine study, it is vital that the background rates of pregnancy and neonatal outcomes are clearly documented as these vary by setting, so that safety signals during vaccine trials can be correctly assessed . Given the important contribution that maternal immunisations could make to reducing maternal and neonatal morbidity, efforts are underway to standardise case definitions used to classify adverse events in maternal vaccine trials. Historically, this has not been the case, limiting comparability between countries and pre and post-licensure. In 2014, in response to a call from the World Health Organisation (WHO) and with funding from the Bill & Melinda Gates Foundation, the GAIA (Global Alignment on Immunisation Safety Assessment in pregnancy) consortium was formed, with the goal of developing a harmonised, globally concerted approach to actively monitor the safety of clinical trials, vaccines and immunization programs in pregnancy. The group have developed 21 standardised case definitions for the classification of adverse obstetric and neonatal events including the need to follow up vaccinated women for 6 months and infants for one year following vaccination.

Study Setting Uganda has a long history of conducting prevention of mother to child HIV transmission (PMTCT) trials as well as vaccine trials for Ebola and Human Immunodeficiency Virus 9. The established National Drug Authority (NDA) and National Immunisation Technical Advisory Group (NITAG) provide pharmacovigilance capacity and an effective platform for monitoring drug and vaccine safety. Makerere University John Hopkins University Research Collaboration (MUJHU) has led multiple PMTCT and HIV therapeutic trials 10. This collaboration with St George's University, who are leaders in immunisation research, presents a unique opportunity to develop a maternal vaccination platform for future trials in Uganda.

Funding has been provided from the European Developing Countries Clinical Trials Partnership (EDCTP) to develop a maternal vaccine trial platform at Kawempe National Referral Hospital. It is anticipated that a tetanus, diptheria and acellular pertussis (Tdap) study will be conducted in 2020 followed by two GBS vaccine trials.

The study site, Kawempe National Referral Hospital, is developing as a centre of excellence for maternal and child health studies in Uganda with several large studies of neonatal encephalopathy, neonatal resuscitation (Clinical Trials - NCT03133572) and birth defects 11 being conducted at the site. Capacity building activities in Kawempe have included implementation and piloting of an electronic medical record (EMR) system to enhance routine data collection. This system provides an opportunity for embedding vaccine surveillance activities for adverse pregnancy outcomes into routine data capture systems which support clinical care.

Kawempe Electronic Medical Record The Uganda Electronic Medical Record (UgandaEMR) is an electronic health record system developed to capture patient level data collected during service delivery. The system is supported by Uganda's Ministry of Health through its Department of Health Informatics (DHI) with technical support from the CDC funded Monitoring and Evaluation Technical support program (METs) under the Makerere University School of Public Health. The system was developed based on open source technology, OpenMRS, and was initially implemented to capture patient level data for HIV care and treatment programs. The system has been rolled out to more than 600 health facilities countrywide and METS aim to rollout it out to 1000 health facilities by the end of 2019. Makerere University John's Hopkins University Research Collaboration (MUJHU) pioneered extension of the system to capture Maternal and Child Health (MCH) information through a pilot implementation initiated in February 2017 in the high-volume national referral hospital in Kawempe, Kampala. Additional data entrants were deployed to capture the e-data in parallel to the standard paper register-based data collection coupled with training and continuous quality improvement measures to support and promote complete and accurate recording in the hospital source forms. An evaluation of the pilot implementation found significant improvement in completeness of both paper and electronic data collected during service delivery from an average of 60% at baseline to over 90% at the end of the pilot implementation period.

GBS Vaccine Research The PREPARE project is an international collaboration that aims to accelerate GBS vaccine development and licensure. It is composed of five work packages (WP). As part of the EDCTP funded PREPARE project two GBS vaccine trials (PREPARE WP4 and 5) will be conducted at Kawempe National Referral Hospital.

In preparation for GBS clinical trials, PREPARE WP2 aims to characterise the Kawempe National Referral hospital baseline pregnancy, neonatal and infant outcomes in preparation for future GBS vaccine trial studies. Pregnancy is associated with complications which must be differentiated from adverse events associated with the administration of vaccines. The frequency of such pregnancy related complications varies significantly by geographical location and the prevalence of such pregnancy and neonatal outcomes are poorly documented in majority of developing countries.

ELIGIBILITY:
Inclusion criteria (Cohort Study):

1. Willing and able to give written informed consent
2. ≥ 14 years of age
3. Pregnant in the first or second trimester
4. Planning to attend routine antenatal care visits and delivery at Kawempe Hospital
5. Planning to stay within Kampala or nearby Wakiso district until at least 9 months post-delivery
6. Willing to attend immunization visits at 10, 6 weeks and 14 weeks to 9 months' end of follow-up visit at Kawempe Hospital
7. Willing to be contacted by phone and/or be visited at home

Inclusion Criteria (EMR) All women and their infants attending for care at Kawempe Hospital during the two years of the study.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants must be pregnant.
Study Population: The study will enrol pregnant women from the general population who present for antenatal care at Kawempe Hospital and follow them and their liveborn infants for a minimum of 14 weeks postpartum up until a maximum of 9 months.
Sampling Method: Non-Probability Sample
Enrollment: 3423 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Maternal, neonatal and infant mortality - Electronic Medical Records. | 24 months
  To describe the maternal and neonatal mortality (%) using hospital electronic medical records (EMR).
Maternal deaths in a prospective cohort. | 24 months
  To describe proportion (%) of maternal deaths in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Maternal gestational diabetes mellitus | 24 months
  To describe proportion (%) of women diagnosed with gestational diabetes mellitus in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Spontaneous abortions & ectopic pregnancy | 24 months
  To describe proportion (%) of women that experience spontaneous abortions and ectopic pregnancies in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Hypertensive disorders | 24 months
  To describe proportion (%) of women that experience hypertensive disorders of pregnancy in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Chorioamnionitis & endometritis | 24 months
  To describe proportion (%) of women that experience chorioamnionitis, endometritis or infection following incomplete abortion in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Haemorrhage | 24 months
  To describe proportion (%) of women that experience antepartum or postpartum haemorrhage in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Fetal distress and dysfunctional labor | 24 months
  To describe proportion (%) of women that experience fetal distress or dysfunctional labor in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Fetal growth restriction | 24 months
  To describe proportion (%) of pregnancies diagnosed with fetal growth restriction in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Birth outcomes (low-birthweight, stillbirths, prematurity) | 24 months
  To describe proportion (%) of births that are low-birthweight, premature or stillborn in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Neonatal outcomes | 24 months
  To describe proportion (%) of liveborn babies that are diagnosed with neonatal encephalopathy, neonatal infections, respiratory distress, seizures or die in the neonatal period in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.
Infant Outcomes | 24 months
  To describe proportion (%) of liveborn babies that die in infancy in a prospective cohort of 4000 mother infant dyads using standardised Global Alignment of Immunisation Safety Assessment in Pregnancy (GAIA) definitions.

SECONDARY OUTCOMES:
Maternal, obstetric, neonatal and infant outcomes - Electronic Medical Records | 24 months
  To describe baseline maternal and neonatal outcomes (as described in the primary objectives) using standards set in the obstetric unit at Kawempe Hospital and GAIA definitions using anonymised data collected using the routine Kawempe electronic medical records (EMR) system.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Le Doare, Dr, Principal Investigator — St George's, University of London
Locations (1):
- MUJHU Care Ltd, Kampala, Uganda

REFERENCES:
- See also: PREPARE Study Website — https://gbsprepare.org